CLINICAL TRIAL: NCT00555204
Title: A Randomized, Double-Blind, Placebo-Controlled Study Using a Bayesian Adaptive Design to Evaluate the Efficacy and Safety of ABT-089 in Subjects With Mild-to-Moderate Alzheimer's Disease on Stable Doses of Acetylcholinesterase Inhibitors
Brief Title: Safety and Efficacy Study of ABT-089 in Adults With Mild to Moderate Alzheimer's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M06-876
Record Dates: First submitted 2007-11-07; First posted 2007-11-08 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Alzheimer's Disease
Keywords: mild to moderate Alzheimer's disease, memory, cognition, dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — pozanicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- A (Experimental)
  Interventions: Drug: ABT-089
- B (Experimental)
  Interventions: Drug: ABT-089
- C (Experimental)
  Interventions: Drug: ABT-089
- D (Experimental)
  Interventions: Drug: ABT-089
- E (Experimental)
  Interventions: Drug: ABT-089
- F (Experimental)
  Interventions: Drug: ABT-089
- G (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ABT-089 — 10 mg - capsules once daily for 12 weeks
  Arms: B
Drug: ABT-089 — 5 mg - capsules once daily for 12 weeks
  Arms: A
Drug: ABT-089 — 15 mg - capsules once daily for 12 weeks
  Arms: C
Drug: ABT-089 — 20 mg - capsules once daily for 12 weeks
  Arms: D
Drug: ABT-089 — 30 mg - capsules once daily for 12 weeks
  Arms: E
Drug: ABT-089 — 35 mg - capsules once daily for 12 weeks
  Arms: F
Drug: placebo — placebo - capsules once daily for 12 weeks
  Arms: G

SUMMARY:
The purpose of this study is to test if the investigational medication ABT-089 is a safe and effective treatment for Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Patient has mild to moderate Alzheimer's disease
* Patient has been receiving a stable dose of an acetylcholinesterase inhibitor
* Patient has a MMSE score between 12 and 26
* Patient has a MHIS score of less than or equal to 4
* Females must be postmenopausal for at least two years or surgically sterile
* Patient has an identified, reliable, caregiver who will support him/her to ensure compliance with treatment and will accompany them to each outpatient visit

Exclusion Criteria:

* Patient is living in a nursing home
* Patient has a history of any significant neurologic disease other than Alzheimer's disease
* Patient has any uncontrolled medical illness
* Patient uses non-prescribed drugs of abuse or has a history of drug or alcohol abuse/dependence

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2007-11; Primary Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | Baseline to Final Evaluation

SECONDARY OUTCOMES:
Pharmacokinetics (how the body handles the study drug) | Baseline to Final Evaluation
Pharmacodynamic (how the study drug affects cognitive functions such as thinking and memory) | Baseline to Final Evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lenz, MD, PhD, Study Director — Abbott
Locations (41):
- United States (41):
  - Phoenix, Arizona
  - Sun City, Arizona
  - Fresno, California
  - San Diego, California
  - Santa Ana, California
  - Santa Monica, California
  - Hamden, Connecticut
  - New Haven, Connecticut
  - Brooksville, Florida
  - Delray Beach, Florida
  - Fort Myers, Florida
  - Hallendale, Florida
  - Hialeah, Florida
  - Largo, Florida
  - Miami, Florida
  - Palm Beach Gardens, Florida
  - Sunrise, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Indianapolis, Indiana
  - Paducah, Kentucky
  - Pittsfield, Massachusetts
  - Grand Rapids, Michigan
  - St Louis, Missouri
  - Long Branch, New Jersey
  - Nutley, New Jersey
  - Princeton, New Jersey
  - Ridgewood, New Jersey
  - Albany, New York
  - New York, New York
  - Staten Island, New York
  - The Bronx, New York
  - Hickory, North Carolina
  - Winston-Salem, North Carolina
  - Centerville, Ohio
  - Cleveland, Ohio
  - Jenkintown, Pennsylvania
  - Norristown, Pennsylvania
  - San Antonio, Texas
  - Wichita Falls, Texas
  - Bennington, Vermont

REFERENCES:
- [Derived] Lenz RA, Pritchett YL, Berry SM, Llano DA, Han S, Berry DA, Sadowsky CH, Abi-Saab WM, Saltarelli MD. Adaptive, dose-finding phase 2 trial evaluating the safety and efficacy of ABT-089 in mild to moderate Alzheimer disease. Alzheimer Dis Assoc Disord. 2015 Jul-Sep;29(3):192-9. doi: 10.1097/WAD.0000000000000093. PMID 25973909